CLINICAL TRIAL: NCT00927277
Title: Erchonia Medical, Inc., Erchonia EML Laser Liposuction Clinical Study V Protocol
Brief Title: Low Level Laser Light Therapy as an Aid to Liposuction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Mr. Steven Shanks, President, Erchonia Medical, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ELIPO-001
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo laser (Placebo Comparator): inactive light on the laser device.
  Interventions: Device: Erchonia(R) LipoLASER PL
- Erchonia (R) LipoLASER PL (Active Comparator): The Erchonia(R) LipoLASER PL is a low level laser light therapy medical device that was applied during the liposuction procedure, by emitting 1 mw of red (635nm wavelength) light via a Class II electric laser diode energy source (CDRH classification). The fluence is considered to be at 10.8 joules per area treated.
  Interventions: Device: Erchonia(R) LipoLASER PL; Erchonia(R) EML Laser

INTERVENTIONS:
Device: Erchonia(R) LipoLASER PL; Erchonia(R) EML Laser — The Erchonia(R) EML Laser is a low level laser light therapy medical device that was applied during the liposuction procedure, by emitting 1 mw of red (635nm wavelength) light via a Class II electric laser diode energy source (CDRH classification). The fluence is considered to be at 10.8 joules per area treated.
  Arms: Erchonia (R) LipoLASER PL
Device: Erchonia(R) LipoLASER PL
  Arms: placebo laser

SUMMARY:
The purpose of this study is to determine whether low level laser therapy can help the recovery process for the procedure of liposuction of the thighs, hips and stomach.

DETAILED DESCRIPTION:
The Erchonia EML Laser is designed to administer low level laser therapy (LLLT). It has been hypothesized that LLLT may reduce pain and promote nerve regeneration through the speculated anti-inflammatory and immune enhancement properties of the therapy. Prior research has indicated LLLT to be a potentially safe and effective means of reducing pain. This clinical study was designed to evaluate the potential of the Erchonia EML Laser in offering a novel means of delivering LLLT to reduce pain and enhance healing following liposuction.

ELIGIBILITY:
Inclusion Criteria: There were separate inclusion criteria for both the liposuction and the clinical study components of the study.

INCLUSION CRITERIA FOR THE LIPOSUCTION PROCEDURE

Prior to partaking in the clinical study qualification evaluation, an individual must have already:

* qualified as a patient for liposuction according to the American Society of Liposuction Surgery (ASLSS) and the American Academy of Cosmetic Surgery (AACS) 2000 Liposuction Guidelines.
* been deemed suitable for undergoing anesthesia according to the American Society of Anesthesiologists: Preanesthesia Evaluation guidelines: Basic Standards For Preanesthesia Care (Approved by House of Delegates on October 14, 1987).
* Signed the physician's standard informed consent form for the liposuction procedure itself.

INCLUSION CRITERIA FOR THE CLINICAL STUDY

* Signed clinical study informed consent form.
* Liposuction procedure intended for the removal of localized deposits of adipose tissue for the purpose of body contouring.
* Body Mass Index (BMI) in kg/m2 of less than 30 (non-obese).
* Localized areas of protruding fat deemed suitable for body contouring liposuction according to the investigator's professional training and experience as for a patient presenting with the same profile and not being considered for participation in the study.
* Areas of treatment to include only one or more of the right and/or left sides of the stomach, thigh, and hips.
* 'Overall firm elastic skin,' as defined by passing of the "snap test" for each intended treatment area.
* American Society of Anesthesiology (ASA) Physical Status Classification System rating of P1: a normal healthy patient or P2: a patient with mild systemic disease, as determined by standard physical examination.
* Suitable for general intubation anesthesia.
* 18 to 55 years, inclusive.

EXCLUSION CRITERIA

* Liposuction procedure intended for the treatment of diseases, such as lipomas, gynecomastia, pseudogynecomastia, lipodystrophy and axillary hyperhydrosis; for the reconstruction of the skin and subtissues in flap elevations, subcutaneous debulking, flap movement or other conditions; to obtain fat for fat transfer (for such purposes as augmentation, correction of scar defects, etc.), and for weight loss.
* ASA Physical Status Classification System rating of P3 to P5.
* Use of narcotics, opiates, steroids and/or NSAIDs within one week prior to surgery.
* Any prior surgery to any of the area(s) to receive liposuction.
* Active infection or wound in any part of the body, including the intended areas of treatment.
* Arthritis or other disorders or injury that directly affect the areas to be treated, including any implants such as pins.
* History of thrombotic events.
* History of neurologic disorder e.g. sensory loss or dysthesia in any of the area(s) to be treated.
* Diabetes.
* Immuno-compromised state, e.g., HIV infection, radiation, chemo or other cancer therapy within the last 6 months.
* Potential bleeding tendencies due to the use of aspirin, non-steroidal anti-inflammatory drugs, estrogen, Vitamin E, herbal supplements such as ginseng, ginger.
* Potential hypercoagulability, e.g., tamoxifen therapy, cancer, recent significant trauma, dehydration.
* Developmental disabilities that affect the ability to read and/or understand the consent form and any other information that may be required from the subject.
* Significant psychological disorder(s) for which treatment has become necessary, including anxiety and depression; psychiatric hospitalization.
* Pregnancy or lactation.
* Involvement in litigation and/or receiving disability benefits related to any kind of disability, injury, or other problem in any one or more of the area(s) to receive liposuction.
* Participation in research during the prior 90 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2003-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Subject self-reported Degree of Pain rating on the standardized 0-100 Visual Analogue Scale (VAS) at 24 hours post-surgery. | 24 hours

SECONDARY OUTCOMES:
Ease of the process of fat extraction during the liposuction procedure | immediately post surgery
Emulsification (consistency) of extracted fat | immediately post surgery
Amount of time spent by volume of fat removed | Immediately post surgery
Degree of swelling at the surgical site | 7 days post surgery
Subject self-reported degree of post-surgical pain | 7, 14 and 28 days post surgery
Use of recovery pain medication | Through the 1st 7 post-surgical days

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Jackson, MD, FACS, Principal Investigator; Gregory Roche, DO, Principal Investigator; Kimberly Butterwick, MD, Principal Investigator

REFERENCES:
- See also: FDA 510(k) clearance listing resulting from the outcome of this clinical study — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=15077